CLINICAL TRIAL: NCT02866227
Title: A Randomized Single Blind Safety and Efficacy Study of TOL-463 Vaginal Gel or Insert in the Treatment of Vaginitis (BV and/or VVC)
Brief Title: TOL-463 Phase 2 Study for Vaginitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Toltec Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-0039; HHSN272201300012I
Record Dates: First submitted 2016-07-28; First posted 2016-08-15 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Bacterial Vaginosis; Vulvovaginal Candidiasis
Keywords: Bacterial; Candidiasis; Gel; Insert; TOL-463; Vaginal; Vaginitis; Vaginoses; Vulvovaginal
MeSH Terms: conditions — Vaginosis, Bacterial; Candidiasis, Vulvovaginal; Candidiasis; Vaginitis | interventions — TOL-463

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BV and/or VVC infection - Gel Treatment (Experimental): Randomized 1:1 to gel nightly for 7 days. N = 40
  Interventions: Drug: TOL-463
- BV and/or VVC infection - Vaginal Insert Treatment (Experimental): Randomized 1:1 to insert nightly for 7 days. N = 40
  Interventions: Drug: TOL-463

INTERVENTIONS:
Drug: TOL-463 — TOL-463 vaginal gel
  Arms: BV and/or VVC infection - Gel Treatment
Drug: TOL-463 — TOL-463 vaginal insert
  Arms: BV and/or VVC infection - Vaginal Insert Treatment

SUMMARY:
This is a Phase II study designed to assess the safety and efficacy of an investigational product, TOL-463, to treat vaginitis.

DETAILED DESCRIPTION:
This is a Phase II randomized single blind safety and efficacy study of TOL-463, administered to female adults to treat vaginitis. Participants will be randomly assigned (1:1) to dose TOL-463 Gel or TOL-463 Insert. Study medication will be administered vaginally, once nightly for seven days. The duration of the study for each participant will be approximately 21-30 days.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible to participate in this study must meet criteria 1 or 2 or both and all of the remaining inclusion criteria:

1. Diagnosis of bacterial vaginosis based on the presence of all four Amsel criteria.*

   * Homogeneous vaginal discharge (off white, milky or gray, thin), positive KOH whiff test, vaginal secretions pH of > 4.5, clue cells > /= 20 percent of vaginal squamous epithelial cells on saline "wet mount"
2. Diagnosis of VVC based on the presence of pseudohyphae on KOH preparation; must also have at least one sign and one symptom*, each rated based on severity** with minimum composite score of 2.

   * Signs include vulvovaginal edema, erythema, and/or excoriation. Symptoms include vulvovaginal itching, burning, and/or irritation. **Severity will be graded on a scale of 0-3 (absent = 0; mild = 1; moderate = 2; severe = 3).
3. Participant is willing and able to provide written informed consent.
4. Participant is 18-50 years of age.
5. Participant is in general good health based on medical history, physical examination, vital signs, and pelvic examination.
6. Any Pap test performed in the prior 3 years must be normal or ASCUS HPV negative.*

   * Consistent with current Pap screening guidelines, a Pap smear must be performed at Visit 1 for any participant who meets the following criteria and cannot provide documentation (which can include self-report) of a normal or ASCUS HPV negative Pap test within the prior 3 years: is 21 years of age or older and (a) has not had a hysterectomy or (b) has had a hysterectomy and has a history of cervical intraepithelial neoplasia grade 2+ (CIN2+) in the past 20 years. If a Pap smear is conducted at Visit 1, the results are not required prior to enrollment.
7. Participant must have a negative urine pregnancy test at study enrollment.
8. Participant must agree to abstain from sexual intercourse during the seven days of study medication use.
9. Participant must be of non-childbearing potential* or must be using highly effective birth control** to avoid becoming pregnant from the time period noted below prior to and through the end of study treatment.

   * Non-childbearing potential is defined as being post-menopausal for at least 1 year, status after bilateral tubal ligation for at least 1 year, or status after bilateral oophorectomy or status after hysterectomy.

     * Acceptable methods of birth control include use of hormonal contraceptives from 30 days prior to study drug dosing or having been abstinent from vaginal sexual intercourse from 21 days prior to study drug dosing and agreeing to abstain from oral, anal, and vaginal sexual intercourse during study drug dosing and, if sexually active, use of non-lubricated condoms (in addition to hormonal contraception) for the remainder of the study through the final visit (V3). Intravaginal or intrauterine contraceptives and contraceptive devices are not acceptable forms of birth control for this study.
10. Participant is willing and able to cooperate to the extent and degree required by this protocol at the discretion of the investigator.
11. Participant is willing to refrain from douching and applying any intravaginal products/medications* throughout the course of the trial.

    * e.g., antifungal preparations, deodorant sprays, spermicides, contraceptive creams, gels, foams, sponges
12. Participant is willing to refrain from using tampons and diaphragms for the seven days of the study product use.

Exclusion Criteria:

1. A diagnosis of vaginitis other than BV or VVC or another vaginal or vulvar condition* that might confuse interpretation of response to study product.

   * Examples of such conditions include erosive lichen planus, desquamative interstitial vaginitis, or contact dermatitis involving the vulvar epithelium.
2. Presence of T. vaginalis on wet mount or evidence of other infectious cause of cervicitis or vaginitis on physical examination.
3. Active genital lesions, including ulcers, vesicles consistent with herpes, or warts.
4. Use of metronidazole or other 5-nitro-imidazole derivative or clindamycin or an antifungal agent (intravaginal or systemic) for the treatment of any condition within 14 days of start of study.
5. Planned ongoing immunosuppressive therapy or systemic antibiotic treatment during the course of the study.
6. Use of any investigational drug within 30 days prior to screening.
7. History of hypersensitivity to any ingredient in the formulations.
8. Women with cervical intraepithelial neoplasia (CIN) or cervical carcinoma.
9. Currently breastfeeding.
10. Menstruating at the time of diagnosis.*

    * Women menstruating at the time of diagnosis may be rescreened at a later time.
11. Any other condition that, in the opinion of the investigator, would interfere with participation in the study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 106 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2017-06-10 (Actual); Study Completion 2017-06-10 (Actual)

PRIMARY OUTCOMES:
Proportion of participants w/ clinical cure (score 0 at TOC for any sign/symptom scored 1-2 at baseline or score 0-1 at TOC for any sign/symptom scored 3 at baseline w/o further treatment needed) at Visit 2 among participants w/ VVC at baseline overall. | Day 9-12
Proportion of participants with clinical cure (defined as absence of: positive KOH whiff test, homogeneous discharge characteristic of BV, clue cells > /= 20% of vaginal squamous epithelial cells) at Visit2 among participants with BV at baseline overall. | Day 9-12
Proportion of participants with clinical cure at Visit 2 among participants with BV at baseline who received TOL-463 Gel. | Day 9-12
Proportion of participants with clinical cure at Visit 2 among participants with BV at baseline who received TOL-463 Insert. | Day 9-12
Proportion of participants with clinical cure at Visit 2 among participants with VVC at baseline who received TOL-463 Gel. | Day 9-12
Proportion of participants with clinical cure at Visit 2 among participants with VVC at baseline who received TOL-463 Insert. | Day 9-12

SECONDARY OUTCOMES:
Among participants with concomitant BV and VVC infections at baseline, the proportion of participants meeting BV clinical cure at Visit 2. | Day 9-12
Among participants with concomitant BV and VVC infections at baseline, the proportion of participants meeting VVC clinical cure at Visit 2. | Day 9-12
The median time (time defined as earliest time point of reported symptom resolution) to symptom relief (at least one day free of all symptoms) as assessed by the participant. | Day 1-7
The occurrence of adverse events considered product-related following initiation of study treatment and through the final study visit. | Day 1-30
The occurrence of secondary VVC following initiation of study treatment and through the final study visit in participants with BV at baseline. | Day 1-30
The proportion of participants experiencing symptom relief (at least one day free of all symptoms) as assessed by the participant. | Day 1-7
The proportion of participants who need additional treatment per physician opinion following initiation of study treatment and through the final study visit. | Day 1-30
The proportion of participants with clinical cure at Visit 3 among participants with BV at baseline. | Day 21-30
The proportion of participants with clinical cure at Visit 3 among participants with VVC at baseline. | Day 21-30
The proportion of participants with microbiologic cure (Nugent score of 0-3) at Visits 2 and 3 among participants with BV at baseline. | Day 9-12, Day 21-30
The proportion of participants with mycological cure at Visits 2 and 3 among participants with VVC at baseline. | Day 9-12, Day 21-30
The proportion of participants with therapeutic cure at Visits 2 and 3 among participants with BV at baseline. | Day 9-12, Day 21-30
The proportion of participants with therapeutic cure at Visits 2 and 3 among participants with VVC at baseline. | Day 9-12, Day 21-30

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama at Birmingham School of Medicine- Infectious Disease, Birmingham, Alabama
  - University of Washington - Harborview Medical Center - Center for AIDS and STD, Seattle, Washington

REFERENCES:
- [Derived] Marrazzo JM, Dombrowski JC, Wierzbicki MR, Perlowski C, Pontius A, Dithmer D, Schwebke J. Safety and Efficacy of a Novel Vaginal Anti-infective, TOL-463, in the Treatment of Bacterial Vaginosis and Vulvovaginal Candidiasis: A Randomized, Single-blind, Phase 2, Controlled Trial. Clin Infect Dis. 2019 Feb 15;68(5):803-809. doi: 10.1093/cid/ciy554. PMID 30184181